CLINICAL TRIAL: NCT06496425
Title: Inspiring Seniors Towards Exercise Promotion to Protect Cognition
Acronym: iSTEP+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Alzheimer's Association (Other); University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Kyoung Shin Park, PhD, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00008531; AARF-23-1145107 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2024-06-12; First posted 2024-07-11 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Physical Activity
Keywords: music; aerobic exercise; strength training; cognition; physical activity; muscular strength; memory complaint
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and music (Experimental): The strength training (ST) program incorporates single-leg exercises for balance training and training with resistance bands and body weight. During the ST, participants will be asked to synchronize their concentric and eccentric muscle contractions in time with the tempo of BMS playlists at a specific music tempo. For aerobic exercise (AE), participants will be instructed to walk at moderate intensity with duration increasing up to an ultimate goal of 150 min/week. Participants will be trained to walk in synchrony with the beats. Participants will receive individualized music playlists to match individual walking cadence and music preference.
  Interventions: Behavioral: Music
- Exercise (No Intervention): The ST program incorporates single-leg exercises for balance training and training with resistance bands and body weight. For AE, participants will be instructed to walk at moderate intensity with duration increasing up to an ultimate goal of 150 min/week.

INTERVENTIONS:
Behavioral: Music — Those randomized to the exercise and music group will receive pre-recorded music playlists along with the exercise. During the strength training (ST), participants will be asked to sync their concentric and eccentric muscle contractions in time with the tempo of playlists. For aerobic exercise (AE), we will adjust the tempo of playlists to match individual walking cadence for participants to be trained to walk in sync with the beats of the playlists.
  Arms: Exercise and music

SUMMARY:
The goal of this clinical trial is to test the benefits of beat-accented music stimulation (BMS) for behavioral changes of physical activity (PA) in older adults with subjective memory complaints. Specific Aims are to determine (1) whether BMS beneficially influences PA behaviors and psychological responses to PA in older adults for 6 months, and (2) whether exercising with BMS differently influences physical and cognitive functioning as well as quality of life in older adults.To test the effects of BMS on PA, participants will be randomly assigned to an exercise intervention that either includes BMS or does not include BMS. Participants will attend a supervised group strength training (ST) (30 min/day) and and aerobic exercise (AE) (30-50 min/day) session for 3 days/week for the first 2 months, 1 day/week for the next 2 months (while encouraging participants to independently perform both AE and ST on other days), and independently for the final 2 months (always with a goal of performing >150min/week AE and 3 days/week of ST for 30 min/day).

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 65 years old.
* Ambulatory/capable of walking for 6 minutes without pain or aid such as a walker/cane.
* Able to speak and read English.
* Healthy enough to exercise at moderate intensity with or without medical clearance by a primary care physician.
* Living in the community for the duration of the study (6 months).
* Having a reliable means of transportation.
* Having a safe place (at least 6 feet by 6 feet of open space) at home for unsupervised exercise training.
* Having self-perceived memory complaints.
* Having no symptoms of suicidal ideation and not meeting criteria for depressive disorder.
* Physically low-active by doing < 60 min/week of moderate-intensity aerobic exercise and no strength training for the last 3 months.

Exclusion Criteria:

* Diagnosis of neurological disorder or spinal cord disorder.
* Known exercise contraindications.
* Current cancer treatment.
* Stroke or neural impairment in the past 6 months.
* Hip/knee/spinal fracture or surgery in the past 6 month.
* Unable or unwilling to attend intervention classes 3x/week in Months 1-2 and 1x/week in Months 3-4.
* Currently participating in any other physical activity or fitness-related research study.
* Use of medication for Alzheimer's disease. Change in dosage of medications prescribed for anxiety or depression within the previous 6 months.
* Regularly drink > 14 alcoholic beverages a week or current illicit drug use.
* Meet the threshold for cognitive impairment.
* Meet the threshold for clinical depression.
* Uncorrected hearing or visual impairments.
* Unable to understand the study procedures.
* One of the household members is participating in this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Changes of physical activity behaviors as assessed by ActiGraph wGT3X-BT | 7 consecutive days at Baseline (before the intervention) and during month 1, 2, 3, 4, 5, and 6
  Duration, intensity, and frequency of physical activity assessed using an waist-worn accelerometer
Affective responses to physical activity as assessed by Physical Activity Enjoyment Scale | At baseline (before the intervention), month 3 and month 5 during the intervention, and post-test (within 4 weeks after the intervention)
  Self-reported affective states relative to physical activity. Physical Activity Enjoyment Scale has 18 items based on a 7-point Likert scale and the total score is ranged from 18 to 126.
Adherence to the physical activity program | A daily exercise log for the entire 6-month period
  Daily duration of aerobic exercise and strength training is self-reported on an exercise log.

SECONDARY OUTCOMES:
General cognition as assessed using the Montreal Cognitive Assessment | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  Montreal Cognitive Assessment takes approximately 10 minutes for completion and the total score is ranged from 0 to 30.
Executive function as assessed using the Tower of London - Freiburg version | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  Tower of London - Freiburg version takes approximately 14 minutes to complete and measures the total number of items solved in minimum number of moves in the range from 0 to 12.
Executive function as assessed using the NIH Toolbox Flanker Inhibitory Control and Attention test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The Flanker Inhibitory Control and Attention test takes approximately 5 minutes to complete and measures the accuracy and reaction time to create a composite score, ranging from 0 to 10.
Executive function as assessed using the NIH Toolbox Dimensional Change Card Sort test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The Dimensional Change Card Sort test takes approximately 5 minutes to complete and measures the accuracy and reaction time to create a composite score, ranging from 0 to 10.
Executive function as assessed using the NIH Toolbox List Sorting Working Memory test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The List Sorting Working Memory test takes approximately 10 minutes to complete and measures the total number of items correctly recalled and sequenced, ranging from 0 to 26.
Episodic memory as assessed using the NIH Toolbox Picture Sequence Memory test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The Picture Sequence Memory test takes approximately 7 minutes to complete and measures the total number of items correctly placed, ranging from 0 to 31, and the IRT-based theta score, ranging from 200 to 700.
Episodic memory as assessed using the Mnemonic Similarity Task | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  This custom-developed test takes approximately 15 minutes to complete and measures mnemonic discrimination (a score ranging from 0-1) and visual recognition (a score ranging from 0-1).
Health-related quality of life as assessed using the RAND 36-Item Short-Form Health Survey | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The RAND 36-Item Short-Form Health Survey Scale has 36 items for self-report, takes 10-15 minutes to complete, and measures health-related quality of life with a score ranging from 0 - 100.
Physical activity behaviors as assessed by physical activity and sedentary behaviour questionnaire. | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The physical activity and sedentary behaviour questionnaire has 7 items and takes approximately 5 minutes for completion
The progress of aerobic capacity and endurance as assessed by 6-minute walk test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
The progress of balance, sit-to-stand, and walking as assessed by Timed Up and Go test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The time taken to complete a Timed Up and Go test is an indicator of fall risks.
The progress of lower-body strength as assessed by 30-Second Sit-to-Stand test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The number of sit-to-stand maneuvers completed in 30 seconds.
The progress of upper-body strength as assessed by Grip Strength test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The squeeze power in pounds measured by by a handheld dynamometer
The progress of balance as assessed by 4-Stage Balance Test | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  The duration of maintaining 4 difference postures
Individual differences in music-related reward experiences as assessed by the Barcelona Music Reward Questionnaire (BMRQ) | At pre-test (before the intervention) and post-test (within 4 weeks after the intervention).
  BMRQ has 24 items and takes 5-10 minutes to complete and measures music-related reward experiences with a score ranging from 0 to 100.
Treatment satisfaction as assessed by the Client Satisfaction Questionnaire (CSQ-8) | At post-test (within 4 weeks after the intervention).
  CSQ has 8 items and takes approximately 3 minutes to complete and measures self-reported satisfaction with the program with a score ranging from 0 to 32.

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Shin Park, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - UNC Greensboro, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park KS, Williams DM, Etnier JL. Exploring the use of music to promote physical activity: From the viewpoint of psychological hedonism. Front Psychol. 2023 Jan 25;14:1021825. doi: 10.3389/fpsyg.2023.1021825. eCollection 2023. PMID 36760458